CLINICAL TRIAL: NCT04146909
Title: The Effect of Lactation on Insulin Sensitivity and Lipolysis in Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study could not be completed as planned due to difficulty to recruit moms during COVID.
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000025731; 1R21HD100751-01 (NIH)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: GDM; Lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast Feeding (Active Comparator): This group will consist of women who exclusively or mostly breast-fed for at least 4-6 months (< 6 ounces of formula/24 hours at 6-9 weeks of delivery)1 and who delivered within the past 18 months.
  Interventions: Diagnostic Test: Hyperinsulinemic-euglycemic clamp
- Formula Feeding (Active Comparator): This group will consist of women who exclusively or mostly formula-fed (no breastfeeding or < 3 weeks of breastfeeding)1 and who delivered within the past 18 months.
  Interventions: Diagnostic Test: Hyperinsulinemic-euglycemic clamp

INTERVENTIONS:
Diagnostic Test: Hyperinsulinemic-euglycemic clamp — After an overnight fast and an equilibration period lasting 2 hours, the 2-step euglycemic-hyperinsulinemic clamp study will be performed. A primed-continuous infusion of regular insulin will be given at 8 mU/(m2 × min) during the first 2 hours, and increased to 40 mU/(m2 × min) for the subsequent 2 hours. Plasma glucose levels will be measured every 5 min, and a variable glucose infusion will be initiated to maintain levels at ∼90 mg/dl. Plasma samples will be drawn at baseline and throughout the infusion period for measurement of isotope enrichment, insulin, NEFA, glycerol turnover, and additional hormones which may be altered with lactation. Approximately 160 mL of blood will be drawn at this visit.

SUMMARY:
This purpose of this study is to investigate whether lactation improves insulin sensitivity and increases lipolysis in women.

DETAILED DESCRIPTION:
There are two aims that this research will address.

In Aim 1, the research question is "Does lactation improve insulin sensitivity and increase lipolysis in women?" In this Aim, researchers will assess whether lactation amongst women with a history of gestational diabetes mellitus (GDM) will improve whole body insulin sensitivity as well as increase whole body lipid turnover by using hyperinsulinemic-euglycemic clamps combined with [6,6-2H]-glucose and [2H5]-glycerol infusions. These stable, non-radiating isotopes have been used extensively and safely to study the mechanisms of insulin resistance amongst non-pregnant as well as pregnant humans; however, these techniques have not previously been applied to the study of insulin sensitivity during lactation. Therefore, the goals will be two-fold: 1) to determine whether lactation induces similar changes in insulin sensitivity in humans as in mice and 2) to pilot the feasibility of performing larger, more detailed metabolic studies in this population of women post-partum.

The second aim (Aim 2) will use a retrospective chart review of women with a history of GDM who had an oral glucose tolerance test (OGTT) 6-8 weeks post-partum as part of standard of care.

The focus of this protocol registration will be Aim 1.

ELIGIBILITY:
Inclusion Criteria:

* A history of GDM (as defined as the American Diabetes Association criteria)
* Delivered a singleton, live birth at ≥ 35 weeks gestation within the past 18 months
* HbA1C < 6.5% at time of screening
* Delivery within the past 18 months
* Breast Feed Group: exclusively or mostly breast-fed (< 6 ounces of formula/24 hours at 6-9 weeks of delivery) for at least 4-6 months

Exclusion Criteria:

* Currently lactating or lactation within the past 1 month at the time of the screening visit
* Diagnosis of diabetes (T1D or T2D) prior to pregnancy
* Current use of any glucose-lowering agents
* Pregnancy related medical problems including preeclampsia
* Major congenital fetal anomalies
* Creatinine > 1.5mg/dL, Hematocrit < 35%, ALT and AST > 2.5X upper limit of normal
* Known psychiatric disorders, alcohol abuse, HIV, hepatitis, renal disease, hepatic disease, untreated heart disease, untreated thyroid disease, active systemic infection or malignancy
* Illicit drug use (by the participant's self-report)
* History of post-partum depression
* Use of weight loss supplements or dieting 6 months prior to study
* Corticosteroid or opiate use within 6 months of study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renate Belfort De Aguiar, MD, PhD, Principal Investigator — Assistant Professor of Medicine (Endocrinology)
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 participants were screened and consented, 1 participant was screened and consented but did not qualify to be on study, demographics were collected from the 6 qualifying participants, with only 3 of those participants receiving intervention. The study could not be completed as planned due to difficulty to recruit moms during COVID.
Groups:
- Breast Fed and Formula Fed: All participants that were breast or formula feeding
Period: Overall Study
Arm/Group | Breast Fed and Formula Fed
Started | 7
Screened, Consented and Qualified | 6
Received Intervention | 3
Completed | 3
Not Completed | 4
Not completed — Withdrawal by Subject | 3
Not completed — Did not qualify after consented | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics presented here are for the 6 participants that were screened, consented and qualified.
Groups:
- Total: Total of all reporting groups
Arm/Group | Breast Feeding | Formula Feeding | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (1.5) | 33 (1.4) | 35 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 2 | 1 | 3
  Asian | 1 | 1 | 2
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32 (7.9) | 34.8 (2.5) | 32.9 (5.3)
Systolic Blood Pressure (BP) [Mean (Standard Deviation); unit: mmHg] | 117 (19) | 148 (27) | 127 (24)
Diastolic BP [Mean (Standard Deviation); unit: mmHg] | 78 (4) | 81 (4) | 79 (4)
Weight [Mean (Standard Deviation); unit: kg] | 87.8 (26.7) | 88.6 (5.7) | 88.1 (17.1)
Body Fat percentage [Mean (Standard Deviation); unit: percentage of body fat] | 43 (9.2) | 46.8 (3.6) | 44.2 (6.4)
Fat Mass [Mean (Standard Deviation); unit: kilograms] | 45.1 (11.8) | 41.5 (5.9) | 43.9 (8.6)
Fat Free Mass (FFM) [Mean (Standard Deviation); unit: kilograms] | 61.4 (22.9) | 47.1 (0.2) | 56.6 (17.4)
Cholesterol [Mean (Standard Deviation); unit: mg/dL]
  Total Cholesterol | 171.3 (18.9) | 185 (49.5) | 175.8 (27)
  High-Density Lipoprotein (HDL) | 55.8 (9.9) | 42 (11.3) | 51.2 (11.6)
  Low-Density Lipoprotein (LDL) | 104.3 (24.7) | 124.5 (28.9) | 111 (25.3)
  Triglycerides | 57.8 (19.2) | 92.5 (46) | 69.3 (31.1)
Glucose Levels [Mean (Standard Deviation); unit: mg/dL] — Change in glucose from fasting baseline to 1 hour by Oral Glucose Tolerance Test (OGTT)
  mg/dL | 66.3 (9.5) | 101.9 (28.1) | 78.1 (23.1)

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Insulin Sensitivity Measured by the Glucose Infusion Rate
Description: The glucose infusion rate is determined by the amount of 20% dextrose given during the hyperinsulinemic-euglycemic clamp study, necessary to keep blood glucose levels at the target range (90-100 mg/dL). Higher rates of infused dextrose indicates greater sensitivity to infused insulin during the hyperinsulinemic-euglycemic clamp. Women with gestational diabetes are expected to be insulin resistant.
Time Frame: 2 hours and 4 hours
Population: Data presented here is from the 3 participants that came to this appointment.
Measure: Mean (Standard Deviation); unit: mg/kg/min
Arm/Group | Breast Feeding | Formula Feeding
Number analyzed (Participants) | 2 | 1
mg/kg/min
  Glucose Infusion Rate 2 hours | 2.1 (1.2) | 1 (NA) — Standard Deviation is not calculable for 1 participant
  Glucose Infusion Rate 4 hours | 7.1 (2.1) | 2.5 (NA) — Standard Deviation is not calculable for 1 participant

2. Primary Outcome: Endogenous Glucose Production
Description: Determined with [6,6-2H] Glucose tracer given during the hyperinsulinemic-euglycemic clamp study. Lower values of endogenous glucose production indicates greater hepatic insulin sensitivity.
Time Frame: 4 hours
Population: Data not collected due to COVID.
Arm/Group | Breast Feeding | Formula Feeding
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Whole Body Lipid Turnover Rates
Description: Determined with [2H5] Glycerol tracer given during the hyperinsulinemic-euglycemic clamp study. Tracer levels in the plasma determinates how the body uses fat in the blood during the hyperinsulinemic-euglycemic clamp study.
Time Frame: 4 hours
Population: Data not collected due to COVID.
Arm/Group | Breast Feeding | Formula Feeding
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Plasma NEFA
Description: Measurement of non-esterified fatty acids levels in the plasma at fasting and during the hyperinsulinemic-euglycemic clamp study. NEFA levels in the plasma are higher in individuals less sensitive to the effects of insulin.
Time Frame: 4 hours
Population: Data not collected due to COVID.
Arm/Group | Breast Feeding | Formula Feeding
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Triglycerides
Description: Measurement of triglycerides levels in the plasma at fasting and during the hyperinsulinemic-euglycemic clamp study. Triglycerides levels in the plasma are higher in individuals less sensitive to the effects of insulin and with type 2 diabetes.
Time Frame: 4 hours
Population: Data not collected due to COVID.
Arm/Group | Breast Feeding | Formula Feeding
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Insulin Levels
Description: Measurement of insulin levels in the plasma at fasting and during the hyperinsulinemic-euglycemic clamp study. Insulin levels in the plasma are higher in insulin resistant individuals.
Time Frame: 4 hours
Population: Data not collected due to COVID.
Arm/Group | Breast Feeding | Formula Feeding
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 hours
Arm/Group | Breast Feeding | Formula Feeding
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04146909/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT04146909/ICF_001.pdf